CLINICAL TRIAL: NCT04186013
Title: Efficacy of Atezolizumab Concurrent With Radiotherapy in Patients With Muscle-invasive Bladder cáncer (Study ATEZOBLADDERPRESERVE)
Brief Title: Efficacy of Atezolizumab Concurrent With Radiotherapy in Patients With Muscle-invasive Bladder cáncer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Spanish Oncology Genito-Urinary Group (Other)
Collaborators: Roche Farma, S.A (Industry); Dynamic Science S.L. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOGUG-2017-A-IEC(VEJ)-4
Record Dates: First submitted 2019-11-26; First posted 2019-12-04 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental): Atezolizumab 1200 mg intravenous infusion every 3 weeks for a total of 6 doses combined with External Beam Radiation Therapy (EBRT) (dosage: 60 Gy in 30 fractions overs 6 weeks at 2Gy/day)
  Interventions: Drug: Atezolizumab Injection [Tecentriq]; Radiation: External Beam Radiation Therapy (EBRT)

INTERVENTIONS:
Drug: Atezolizumab Injection [Tecentriq] — intravenous infusion of 1.200 mg of Atezolizumab administered intravenously every 3 weeks for a total of 6 doses
Radiation: External Beam Radiation Therapy (EBRT) — 60 Gy of radiotherapy in 30 fractions overs 6 weeks at 2 Gy/day

SUMMARY:
Open, multicentre, phase II trial of atezolizumab with concurrent normofractionated radiotherapy in patients with localized muscle-invasive bladder cancer treated with a selective multimodality bladder conservative approach.

DETAILED DESCRIPTION:
STUDY DESIGN:

Open, multicentre, phase II trial of atezolizumab with concurrent normofractionated radiotherapy in patients with histologically confirmed diagnosis of muscle-invasive urothelial carcinoma of the bladder.

The bladder preserving therapy include combined modality therapy with:

STUDY TREATMENTS:

Investigational product (atezolizumab/Tecentriq ®):

* Route of administration: intravenous infusion.
* Duration of treatment: 16 weeks.
* Dosage: 1.200 mg intravenous every 3 weeks for a total of 6 doses. Atezolizumab is supplied as atezolizumab 1200 mg/20 mL vials (60 mg/mL) solution for intravenous infusion. After dilution, one mL of solution should contain approximately 4.4 mg of atezolizumab (1,200 mg/270 mL).

External Beam Radiation Therapy (EBRT): radiation

* Duration of treatment: 6 weeks
* Dosage: 60 Gy of radiotherapy in 30 fractions overs 6 weeks at 2Gy/day

STUDY POPULATION:

Adult patients (aged ≥18 years) with histologically confirmed diagnosis of muscle-invasive urothelial carcinoma of the bladder, in clinical stages T2-T4a who are not candidates for radical cystectomy by medical reasons, refusal or patient´s choice.

A total of 39 patients are estimated to be included in the study.

OBJECTIVES:

Primary objective:

The primary objective of the study is to determine the efficacy of atezolizumab concurrent with radiotherapy in terms of pathological complete response defined as a response of grade 5 according to Miller and Payne criteria in patients with muscle-invasive bladder cancer treated with bladder preservation intent.

Secondary objectives:

* To evaluate overall survival (OS).
* To evaluate disease specific survival (DSS).
* To evaluate disease free survival (DFS).
* To evaluate bladder intact disease-free survival (BIDFS).
* To calculate the number of patients with muscle invasive and non-muscle invasive local failure (LF).
* To determine the rate of distance metastases defined as the percentage of patients who develop metastases.
* To determine to the rate of patients with bladder preserved.
* To determine to the rate of immediate or late salvage cystectomy.
* The safety profile and tolerability of the combination of atezolizumab with concurrent radiotherapy.

Exploratory objectives:

* To determine the predictive role of the expression of PD-1 / PD-L1 and CD8 in terms of pCR, OS and DFS in bladder cancer patients treated with atezolizumab plus radiotherapy.
* The correlation between the levels of IFN-γ, interleukin 6 (IL-6), interleukin 18 (IL-18), or ITAC (also called CXCL11 or IP-9) and the efficacy parameters (pCR, OS and DFS) of the treatment with atezolizumab plus radiotherapy.

STUDY VISITS AND PROCEDURES:

The study includes the following visits:

* Screening: within the 28 days prior to starting the study treatment.
* Baseline visit: the first day of cycle 1
* Visits over the treatment period (16 weeks ± 7 days): from administration of the first dose of the study treatment to the administration of the last dose of atezolizumab or withdrawal from the treatment. Treatment will consist of the administration of atezolizumab at 1,200 mg intravenous every 3 weeks for 6 cycles
* Post-treatment follow-up: includes the biopsy and safety visit 1-2 months after the last dose of atezolizumab and a subsequent 5 years follow-up period after.
* End of study visit/ Early termination: In patients who end the study follow-up or prematurely withdraw from the study

ELIGIBILITY:
Inclusion criteria:

1. Patients must be 18 years of age or older.
2. Patients have histologically-confirmed diagnosis of muscle-invasive urothelial carcinoma of the bladder, in clinical stages T2-4a N0 M0, who are not candidates for radical cystectomy by medical reasons, refusal or patient's choice.
3. Patients who refuse treatment with cisplatin-based chemotherapy or in whom treatment with cisplatin-based therapy is not appropriate.
4. Patients must have ECOG performance status 0 to 2.
5. Patients must have adequate bone marrow function as defined by absolute neutrophil count >1.500/mm3; platelets >100.000/mm3 and HB ≥ 9g/dl.
6. Patients must have adequate renal and liver function as defined by calculated creatinine clearance >15ml/min.
7. Total bilirubin, SGOT (AST) and/or SGPT (ALT) < 2,5 times the upper limit of normal.
8. International Normalized Ration (INR) or Prothrombin Time (PT): ≤1.5 X ULN unless participant is receiving anticoagulant therapy (as long as PT or PTT is within therapeutic range of intended use of anticoagulants).
9. Activated Partial Thromboplastin Time (aPTT): ≤1.5 X ULN unless participant is receiving anticoagulant therapy (as long as PT or PTT is within therapeutic range of intended use of anticoagulants).
10. Female participant of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to registering the patient. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
11. Female participants of childbearing potential should be willing to use two methods of birth control or be surgically sterile or abstain from heterosexual activity for the course of the study through 5 months after the last dose of study medication. Participants of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
12. Male participants should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy (1).
13. A paraffin-embedded tumour sample must be available for the associate molecular study.

Exclusion criteria:

1. Previous treatment with radiotherapy to the bladder, systemic chemotherapy or immune checkpoint inhibitors. Prior intravesical BCG treatment for non-muscle invasive bladder cancer is allowed.
2. Presence of regional lymph node or metastatic extension of the disease.
3. Concurrent treatment with other experimental drugs (within 30 days prior to study entry) or other anti-cancer therapy.
4. History of prior malignancies within the preceding 5 years other than previously treated basal cell carcinoma of the skin, non-muscle invasive bladder cancer, incidental prostate carcinoma Stage T1a well differentiated prostatic carcinoma in men (Gleason = 3+3, PSA <5) and carcinoma in situ of the cervix.
5. Evidence of tumour-related moderate/severe hydronephrosis unless stented or with nephrostomy to preserve renal function.
6. Extensive or multifocal bladder carcinoma in situ (CIS) precluding curative chemoradiotherapy.
7. Bulky T3/T4a tumours unsuitable for curative treatment (i.e. > 5 cm in any dimension). Tumours measures must be done post-TUR via CT scan.
8. Patients with serious uncontrolled infection.
9. Has a known history of active BT (Bacillus Tuberculosis).
10. Has known history of, or any evidence of active, non-infectious pneumonitis.
11. Autoimmune diseases other than vitiligo, type I diabetes mellitus, residual hypothyroidism requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger.
12. Positive test for hepatitis B virus surface antigen (HBVsAg) or hepatitis C virus ribonucleic acid antibody (HCV-Ab) indicating acute or chronic infection.
13. Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
14. Subjects with a condition requiring systemic treatment with either corticosteroids (equivalent to > 10 mg/day prednisone) or other immune-suppressive medications within 14 days of study drug administration.
15. Women of child-bearing potential unwilling to be abstinent or use effective methods of birth control.
16. General medical or psychological conditions that would preclude appropriate informed consent or compliance with the protocol.

(1) Acceptable methods of effective contraception:

* Complete sexual abstinence for 14 days before the start of study treatment to 5 months after completion of the investigational treatment.
* Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy), or tubal ligation at least six weeks before taking study treatment.
* Male sterilization (at least 6 months prior to screening). For female subjects on the study the vasectomized male partner should be the sole partner for that subject.
* Intrauterine device or system with a documented failure less than 1%.
* Double barrier method with spermicide.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2019-09-18 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response | After the end of the treatment (16 weeks)
  Response of grade 5 according to Miller and Payne criteria

SECONDARY OUTCOMES:
Overall survival | through study completion, up to 5 years
  Time from the date of the beginning of protocol therapy to the date of death due to any cause
Disease specific survival | through study completion, up to 5 years
  Time from start of treatment to the date of having evidence of distant metastases, nodal recurrence or recurrence within the radiotherapy field that could be salvaged in a curative fashion, what happens first
Disease free survival | through study completion, up to 5 years
  Time from the date of start of protocol therapy to the date of recurrence of muscle invasive or non-invasive bladder carcinoma or metastases, what happens first
Bladder-intact disease-free survival | through study completion, up to 5 years
  Time from the date of initiation of protocol therapy until the development of MIBC recurrence, regional pelvic recurrence, distant metastases, bladder cancer-related death or cystectomy, what happens first
Muscle invasive and non-muscle invasive local failure | through study completion, up to 5 years
  defined as patients that do not achieve a pCR defined as a response of grade 5 according to Miller and Payne criteria and documented tumour recurrence after pCR
Rate of distant metastases | through study completion, up to 5 years
  Percentage of patients who develop distant metastases. Defined as lymphonodal involvement above the bifurcation of the iliac vessels or in inquinal regions and metastases resulting from hematogenous spread
Rate of patients with bladder preserved | through study completion, up to 5 years
  Rate of patients with bladder preserved at the time of the biopsy of the tumour performed between one and two months after the last dose of atezolizumab
Rate of immediate or late salvage cystectomy | through study completion, up to 5 years
  Immediate will be evaluated at the time of the biopsy of the tumour performed between one and two months after the last dose of atezolizumab and late will be evaluated during the follow-up
The safety profile and tolerability of the combination of atezolizumab with concurrent radiotherapy | through study completion, up to 5 years
  Collection of any adverse events and serious adverse events

CONTACTS AND LOCATIONS:
Locations (10):
- Spain (10):
  - Althaia Xarxa Assintencial, Manresa, Barcelona
  - Consorci Corporació Sanitària Parc Taulí, Sabadell, Barcelona
  - Hospital Universitario Sant Joan de Reus, Reus, Tarragona
  - Hospital Clínico Universitario San Cecilio, Granada
  - Hospital Universitario Lucus Augusti, Lugo
  - Hospital Universitario La Princesa, Madrid
  - Hospital HM Sanchinarro, Madrid
  - Complejo Hospitalario Universitario Ourense, Ourense
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Arnau de Vilanova, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Torre LA, Bray F, Siegel RL, Ferlay J, Lortet-Tieulent J, Jemal A. Global cancer statistics, 2012. CA Cancer J Clin. 2015 Mar;65(2):87-108. doi: 10.3322/caac.21262. Epub 2015 Feb 4. PMID 25651787
- [Result] Stenzl A, Burger M, Fradet Y, Mynderse LA, Soloway MS, Witjes JA, Kriegmair M, Karl A, Shen Y, Grossman HB. Hexaminolevulinate guided fluorescence cystoscopy reduces recurrence in patients with nonmuscle invasive bladder cancer. J Urol. 2010 Nov;184(5):1907-13. doi: 10.1016/j.juro.2010.06.148. Epub 2010 Sep 17. PMID 20850152
- [Result] Geavlete B, Jecu M, Multescu R, Geavlete P. Narrow-band imaging cystoscopy in non-muscle-invasive bladder cancer: a prospective comparison to the standard approach. Ther Adv Urol. 2012 Oct;4(5):211-7. doi: 10.1177/1756287212454181. PMID 23024703
- [Result] Naselli A, Introini C, Timossi L, Spina B, Fontana V, Pezzi R, Germinale F, Bertolotto F, Puppo P. A randomized prospective trial to assess the impact of transurethral resection in narrow band imaging modality on non-muscle-invasive bladder cancer recurrence. Eur Urol. 2012 May;61(5):908-13. doi: 10.1016/j.eururo.2012.01.018. Epub 2012 Jan 20. PMID 22280855
- [Result] Xiong Y, Li J, Ma S, Ge J, Zhou L, Li D, Chen Q. A meta-analysis of narrow band imaging for the diagnosis and therapeutic outcome of non-muscle invasive bladder cancer. PLoS One. 2017 Feb 13;12(2):e0170819. doi: 10.1371/journal.pone.0170819. eCollection 2017. PMID 28192481
- [Result] Humphrey PA, Moch H, Cubilla AL, Ulbright TM, Reuter VE. The 2016 WHO Classification of Tumours of the Urinary System and Male Genital Organs-Part B: Prostate and Bladder Tumours. Eur Urol. 2016 Jul;70(1):106-119. doi: 10.1016/j.eururo.2016.02.028. Epub 2016 Mar 17. PMID 26996659
- [Result] Murta-Nascimento C, Silverman DT, Kogevinas M, Garcia-Closas M, Rothman N, Tardon A, Garcia-Closas R, Serra C, Carrato A, Villanueva C, Dosemeci M, Real FX, Malats N. Risk of bladder cancer associated with family history of cancer: do low-penetrance polymorphisms account for the increase in risk? Cancer Epidemiol Biomarkers Prev. 2007 Aug;16(8):1595-600. doi: 10.1158/1055-9965.EPI-06-0743. PMID 17684133
- [Result] Ploeg M, Aben KK, Kiemeney LA. The present and future burden of urinary bladder cancer in the world. World J Urol. 2009 Jun;27(3):289-93. doi: 10.1007/s00345-009-0383-3. Epub 2009 Feb 15. PMID 19219610
- [Result] Madersbacher S, Hochreiter W, Burkhard F, Thalmann GN, Danuser H, Markwalder R, Studer UE. Radical cystectomy for bladder cancer today--a homogeneous series without neoadjuvant therapy. J Clin Oncol. 2003 Feb 15;21(4):690-6. doi: 10.1200/JCO.2003.05.101. PMID 12586807
- [Result] Babjuk M, Bohle A, Burger M, Capoun O, Cohen D, Comperat EM, Hernandez V, Kaasinen E, Palou J, Roupret M, van Rhijn BWG, Shariat SF, Soukup V, Sylvester RJ, Zigeuner R. EAU Guidelines on Non-Muscle-invasive Urothelial Carcinoma of the Bladder: Update 2016. Eur Urol. 2017 Mar;71(3):447-461. doi: 10.1016/j.eururo.2016.05.041. Epub 2016 Jun 17. PMID 27324428
- [Result] Arcangeli G, Arcangeli S, Strigari L. A systematic review and meta-analysis of clinical trials of bladder-sparing trimodality treatment for muscle-invasive bladder cancer (MIBC). Crit Rev Oncol Hematol. 2015 Apr;94(1):105-15. doi: 10.1016/j.critrevonc.2014.11.007. Epub 2014 Dec 4. PMID 25541350
- [Result] Efstathiou JA, Spiegel DY, Shipley WU, Heney NM, Kaufman DS, Niemierko A, Coen JJ, Skowronski RY, Paly JJ, McGovern FJ, Zietman AL. Long-term outcomes of selective bladder preservation by combined-modality therapy for invasive bladder cancer: the MGH experience. Eur Urol. 2012 Apr;61(4):705-11. doi: 10.1016/j.eururo.2011.11.010. Epub 2011 Nov 12. PMID 22101114
- [Result] James ND, Hussain SA, Hall E, Jenkins P, Tremlett J, Rawlings C, Crundwell M, Sizer B, Sreenivasan T, Hendron C, Lewis R, Waters R, Huddart RA; BC2001 Investigators. Radiotherapy with or without chemotherapy in muscle-invasive bladder cancer. N Engl J Med. 2012 Apr 19;366(16):1477-88. doi: 10.1056/NEJMoa1106106. PMID 22512481
- [Result] Mak KS, Smith AB, Eidelman A, Clayman R, Niemierko A, Cheng JS, Matthews J, Drumm MR, Nielsen ME, Feldman AS, Lee RJ, Zietman AL, Chen RC, Shipley WU, Milowsky MI, Efstathiou JA. Quality of Life in Long-term Survivors of Muscle-Invasive Bladder Cancer. Int J Radiat Oncol Biol Phys. 2016 Dec 1;96(5):1028-1036. doi: 10.1016/j.ijrobp.2016.08.023. Epub 2016 Aug 24. PMID 27727064
- [Result] Huddart RA, Birtle A, Maynard L, Beresford M, Blazeby J, Donovan J, Kelly JD, Kirkbank T, McLaren DB, Mead G, Moynihan C, Persad R, Scrase C, Lewis R, Hall E. Clinical and patient-reported outcomes of SPARE - a randomised feasibility study of selective bladder preservation versus radical cystectomy. BJU Int. 2017 Nov;120(5):639-650. doi: 10.1111/bju.13900. Epub 2017 May 29. PMID 28453896
- [Result] Gray PJ, Lin CC, Jemal A, Shipley WU, Fedewa SA, Kibel AS, Rosenberg JE, Kamat AM, Virgo KS, Blute ML, Zietman AL, Efstathiou JA. Clinical-pathologic stage discrepancy in bladder cancer patients treated with radical cystectomy: results from the national cancer data base. Int J Radiat Oncol Biol Phys. 2014 Apr 1;88(5):1048-56. doi: 10.1016/j.ijrobp.2014.01.001. PMID 24661658
- [Result] Hagan MP, Winter KA, Kaufman DS, Wajsman Z, Zietman AL, Heney NM, Toonkel LM, Jones CU, Roberts JD, Shipley WU. RTOG 97-06: initial report of a phase I-II trial of selective bladder conservation using TURBT, twice-daily accelerated irradiation sensitized with cisplatin, and adjuvant MCV combination chemotherapy. Int J Radiat Oncol Biol Phys. 2003 Nov 1;57(3):665-72. doi: 10.1016/s0360-3016(03)00718-1. PMID 14529770
- [Result] Rodel C, Grabenbauer GG, Kuhn R, Papadopoulos T, Dunst J, Meyer M, Schrott KM, Sauer R. Combined-modality treatment and selective organ preservation in invasive bladder cancer: long-term results. J Clin Oncol. 2002 Jul 15;20(14):3061-71. doi: 10.1200/JCO.2002.11.027. PMID 12118019
- [Result] Bellmunt J, Theodore C, Demkov T, Komyakov B, Sengelov L, Daugaard G, Caty A, Carles J, Jagiello-Gruszfeld A, Karyakin O, Delgado FM, Hurteloup P, Winquist E, Morsli N, Salhi Y, Culine S, von der Maase H. Phase III trial of vinflunine plus best supportive care compared with best supportive care alone after a platinum-containing regimen in patients with advanced transitional cell carcinoma of the urothelial tract. J Clin Oncol. 2009 Sep 20;27(27):4454-61. doi: 10.1200/JCO.2008.20.5534. Epub 2009 Aug 17. PMID 19687335
- [Result] Zhang S, Yu YH, Zhang Y, Qu W, Li J. Radiotherapy in muscle-invasive bladder cancer: the latest research progress and clinical application. Am J Cancer Res. 2015 Jan 15;5(2):854-68. eCollection 2015. PMID 25973322
- [Result] Baumeister SH, Freeman GJ, Dranoff G, Sharpe AH. Coinhibitory Pathways in Immunotherapy for Cancer. Annu Rev Immunol. 2016 May 20;34:539-73. doi: 10.1146/annurev-immunol-032414-112049. Epub 2016 Feb 25. PMID 26927206
- [Result] Dong H, Strome SE, Salomao DR, Tamura H, Hirano F, Flies DB, Roche PC, Lu J, Zhu G, Tamada K, Lennon VA, Celis E, Chen L. Tumor-associated B7-H1 promotes T-cell apoptosis: a potential mechanism of immune evasion. Nat Med. 2002 Aug;8(8):793-800. doi: 10.1038/nm730. Epub 2002 Jun 24. PMID 12091876
- [Result] Inman BA, Sebo TJ, Frigola X, Dong H, Bergstralh EJ, Frank I, Fradet Y, Lacombe L, Kwon ED. PD-L1 (B7-H1) expression by urothelial carcinoma of the bladder and BCG-induced granulomata: associations with localized stage progression. Cancer. 2007 Apr 15;109(8):1499-505. doi: 10.1002/cncr.22588. PMID 17340590
- [Result] Robert C, Long GV, Brady B, Dutriaux C, Maio M, Mortier L, Hassel JC, Rutkowski P, McNeil C, Kalinka-Warzocha E, Savage KJ, Hernberg MM, Lebbe C, Charles J, Mihalcioiu C, Chiarion-Sileni V, Mauch C, Cognetti F, Arance A, Schmidt H, Schadendorf D, Gogas H, Lundgren-Eriksson L, Horak C, Sharkey B, Waxman IM, Atkinson V, Ascierto PA. Nivolumab in previously untreated melanoma without BRAF mutation. N Engl J Med. 2015 Jan 22;372(4):320-30. doi: 10.1056/NEJMoa1412082. Epub 2014 Nov 16. PMID 25399552
- [Result] Brown JA, Dorfman DM, Ma FR, Sullivan EL, Munoz O, Wood CR, Greenfield EA, Freeman GJ. Blockade of programmed death-1 ligands on dendritic cells enhances T cell activation and cytokine production. J Immunol. 2003 Feb 1;170(3):1257-66. doi: 10.4049/jimmunol.170.3.1257. PMID 12538684
- [Result] Latchman Y, Wood CR, Chernova T, Chaudhary D, Borde M, Chernova I, Iwai Y, Long AJ, Brown JA, Nunes R, Greenfield EA, Bourque K, Boussiotis VA, Carter LL, Carreno BM, Malenkovich N, Nishimura H, Okazaki T, Honjo T, Sharpe AH, Freeman GJ. PD-L2 is a second ligand for PD-1 and inhibits T cell activation. Nat Immunol. 2001 Mar;2(3):261-8. doi: 10.1038/85330. PMID 11224527
- [Result] Boorjian SA, Sheinin Y, Crispen PL, Farmer SA, Lohse CM, Kuntz SM, Leibovich BC, Kwon ED, Frank I. T-cell coregulatory molecule expression in urothelial cell carcinoma: clinicopathologic correlations and association with survival. Clin Cancer Res. 2008 Aug 1;14(15):4800-8. doi: 10.1158/1078-0432.CCR-08-0731. PMID 18676751
- [Result] Topalian SL, Hodi FS, Brahmer JR, Gettinger SN, Smith DC, McDermott DF, Powderly JD, Carvajal RD, Sosman JA, Atkins MB, Leming PD, Spigel DR, Antonia SJ, Horn L, Drake CG, Pardoll DM, Chen L, Sharfman WH, Anders RA, Taube JM, McMiller TL, Xu H, Korman AJ, Jure-Kunkel M, Agrawal S, McDonald D, Kollia GD, Gupta A, Wigginton JM, Sznol M. Safety, activity, and immune correlates of anti-PD-1 antibody in cancer. N Engl J Med. 2012 Jun 28;366(26):2443-54. doi: 10.1056/NEJMoa1200690. Epub 2012 Jun 2. PMID 22658127
- [Result] Patel SP, Kurzrock R. PD-L1 Expression as a Predictive Biomarker in Cancer Immunotherapy. Mol Cancer Ther. 2015 Apr;14(4):847-56. doi: 10.1158/1535-7163.MCT-14-0983. Epub 2015 Feb 18. PMID 25695955
- [Result] Powles T, Eder JP, Fine GD, Braiteh FS, Loriot Y, Cruz C, Bellmunt J, Burris HA, Petrylak DP, Teng SL, Shen X, Boyd Z, Hegde PS, Chen DS, Vogelzang NJ. MPDL3280A (anti-PD-L1) treatment leads to clinical activity in metastatic bladder cancer. Nature. 2014 Nov 27;515(7528):558-62. doi: 10.1038/nature13904. PMID 25428503
- [Result] Herbst RS, Soria JC, Kowanetz M, Fine GD, Hamid O, Gordon MS, Sosman JA, McDermott DF, Powderly JD, Gettinger SN, Kohrt HE, Horn L, Lawrence DP, Rost S, Leabman M, Xiao Y, Mokatrin A, Koeppen H, Hegde PS, Mellman I, Chen DS, Hodi FS. Predictive correlates of response to the anti-PD-L1 antibody MPDL3280A in cancer patients. Nature. 2014 Nov 27;515(7528):563-7. doi: 10.1038/nature14011. PMID 25428504
- [Result] Phillips T, Simmons P, Inzunza HD, Cogswell J, Novotny J Jr, Taylor C, Zhang X. Development of an automated PD-L1 immunohistochemistry (IHC) assay for non-small cell lung cancer. Appl Immunohistochem Mol Morphol. 2015 Sep;23(8):541-9. doi: 10.1097/PAI.0000000000000256. PMID 26317305
- [Result] Zhang X, Schwartz JC, Guo X, Bhatia S, Cao E, Lorenz M, Cammer M, Chen L, Zhang ZY, Edidin MA, Nathenson SG, Almo SC. Structural and functional analysis of the costimulatory receptor programmed death-1. Immunity. 2004 Mar;20(3):337-47. doi: 10.1016/s1074-7613(04)00051-2. PMID 15030777
- [Result] Avci N, Deligonul A, Tolunay S, Cubukcu E, Fatih Olmez O, Altmisdortoglu O, Tanriverdi O, Aksoy A, Kurt E, Evrensel T. Prognostic impact of tumor lymphocytic infiltrates in patients with breast cancer undergoing neoadjuvant chemotherapy. J BUON. 2015 Jul-Aug;20(4):994-1000. PMID 26416041
- [Result] Pham CD, Flores C, Yang C, Pinheiro EM, Yearley JH, Sayour EJ, Pei Y, Moore C, McLendon RE, Huang J, Sampson JH, Wechsler-Reya R, Mitchell DA. Differential Immune Microenvironments and Response to Immune Checkpoint Blockade among Molecular Subtypes of Murine Medulloblastoma. Clin Cancer Res. 2016 Feb 1;22(3):582-95. doi: 10.1158/1078-0432.CCR-15-0713. Epub 2015 Sep 24. PMID 26405194
- [Result] Lemanska-Perek A, Lis-Kuberka J, Lepczynski A, Dratwa-Chalupnik A, Tupikowski K, Katnik-Prastowska I, Ozgo M. Potential plasma biomarkers of bladder cancer identified by proteomic analysis: A pilot study. Adv Clin Exp Med. 2019 Mar;28(3):339-346. doi: 10.17219/acem/79296. PMID 29963784
- [Result] Trinchieri G, Perussia B. Immune interferon: a pleiotropic lymphokine with multiple effects. Immunol Today. 1985 Apr;6(4):131-6. doi: 10.1016/0167-5699(85)90080-5. PMID 25289500
- [Result] Basham TY, Merigan TC. Recombinant interferon-gamma increases HLA-DR synthesis and expression. J Immunol. 1983 Apr;130(4):1492-4. PMID 6403609
- [Result] Ozzello L, Habif DV, De Rosa CM, Cantell K. Cellular events accompanying regression of skin recurrences of breast carcinomas treated with intralesional injections of natural interferons alpha and gamma. Cancer Res. 1992 Sep 1;52(17):4571-81. PMID 1355007
- [Result] Hawkyard SJ, Jackson AM, James K, Prescott S, Smyth JF, Chisholm GD. The inhibitory effects of interferon gamma on the growth of bladder cancer cells. J Urol. 1992 May;147(5):1399-403. doi: 10.1016/s0022-5347(17)37582-1. PMID 1569695
- [Result] Novick D, Engelmann H, Wallach D, Leitner O, Revel M, Rubinstein M. Purification of soluble cytokine receptors from normal human urine by ligand-affinity and immunoaffinity chromatography. J Chromatogr. 1990 Jun 27;510:331-7. doi: 10.1016/s0021-9673(01)93767-7. PMID 2144854
- [Result] Ruckert M, Deloch L, Fietkau R, Frey B, Hecht M, Gaipl US. Immune modulatory effects of radiotherapy as basis for well-reasoned radioimmunotherapies. Strahlenther Onkol. 2018 Jun;194(6):509-519. doi: 10.1007/s00066-018-1287-1. Epub 2018 Mar 2. PMID 29500551
- [Result] Kroemer G, Galluzzi L, Kepp O, Zitvogel L. Immunogenic cell death in cancer therapy. Annu Rev Immunol. 2013;31:51-72. doi: 10.1146/annurev-immunol-032712-100008. Epub 2012 Nov 12. PMID 23157435
- [Result] Sistigu A, Yamazaki T, Vacchelli E, Chaba K, Enot DP, Adam J, Vitale I, Goubar A, Baracco EE, Remedios C, Fend L, Hannani D, Aymeric L, Ma Y, Niso-Santano M, Kepp O, Schultze JL, Tuting T, Belardelli F, Bracci L, La Sorsa V, Ziccheddu G, Sestili P, Urbani F, Delorenzi M, Lacroix-Triki M, Quidville V, Conforti R, Spano JP, Pusztai L, Poirier-Colame V, Delaloge S, Penault-Llorca F, Ladoire S, Arnould L, Cyrta J, Dessoliers MC, Eggermont A, Bianchi ME, Pittet M, Engblom C, Pfirschke C, Preville X, Uze G, Schreiber RD, Chow MT, Smyth MJ, Proietti E, Andre F, Kroemer G, Zitvogel L. Cancer cell-autonomous contribution of type I interferon signaling to the efficacy of chemotherapy. Nat Med. 2014 Nov;20(11):1301-9. doi: 10.1038/nm.3708. Epub 2014 Oct 26. PMID 25344738
- [Result] Chiappinelli KB, Strissel PL, Desrichard A, Li H, Henke C, Akman B, Hein A, Rote NS, Cope LM, Snyder A, Makarov V, Budhu S, Slamon DJ, Wolchok JD, Pardoll DM, Beckmann MW, Zahnow CA, Merghoub T, Chan TA, Baylin SB, Strick R. Inhibiting DNA Methylation Causes an Interferon Response in Cancer via dsRNA Including Endogenous Retroviruses. Cell. 2017 Apr 6;169(2):361. doi: 10.1016/j.cell.2017.03.036. No abstract available. PMID 28388418
- [Result] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Result] Rosenberg JE, Hoffman-Censits J, Powles T, van der Heijden MS, Balar AV, Necchi A, Dawson N, O'Donnell PH, Balmanoukian A, Loriot Y, Srinivas S, Retz MM, Grivas P, Joseph RW, Galsky MD, Fleming MT, Petrylak DP, Perez-Gracia JL, Burris HA, Castellano D, Canil C, Bellmunt J, Bajorin D, Nickles D, Bourgon R, Frampton GM, Cui N, Mariathasan S, Abidoye O, Fine GD, Dreicer R. Atezolizumab in patients with locally advanced and metastatic urothelial carcinoma who have progressed following treatment with platinum-based chemotherapy: a single-arm, multicentre, phase 2 trial. Lancet. 2016 May 7;387(10031):1909-20. doi: 10.1016/S0140-6736(16)00561-4. Epub 2016 Mar 4. PMID 26952546
- [Result] Ahmed KA, Stallworth DG, Kim Y, Johnstone PA, Harrison LB, Caudell JJ, Yu HH, Etame AB, Weber JS, Gibney GT. Clinical outcomes of melanoma brain metastases treated with stereotactic radiation and anti-PD-1 therapy. Ann Oncol. 2016 Mar;27(3):434-41. doi: 10.1093/annonc/mdv622. Epub 2015 Dec 27. PMID 26712903
- [Result] Mayor S. Radiation in combination with immune-checkpoint inhibitors. Lancet Oncol. 2015 Apr;16(4):e162. doi: 10.1016/S1470-2045(15)70118-X. Epub 2015 Mar 13. No abstract available. PMID 25773169
- [Result] Sharabi AB, Lim M, DeWeese TL, Drake CG. Radiation and checkpoint blockade immunotherapy: radiosensitisation and potential mechanisms of synergy. Lancet Oncol. 2015 Oct;16(13):e498-509. doi: 10.1016/S1470-2045(15)00007-8. PMID 26433823
- [Result] Fehrenbacher L, Spira A, Ballinger M, Kowanetz M, Vansteenkiste J, Mazieres J, Park K, Smith D, Artal-Cortes A, Lewanski C, Braiteh F, Waterkamp D, He P, Zou W, Chen DS, Yi J, Sandler A, Rittmeyer A; POPLAR Study Group. Atezolizumab versus docetaxel for patients with previously treated non-small-cell lung cancer (POPLAR): a multicentre, open-label, phase 2 randomised controlled trial. Lancet. 2016 Apr 30;387(10030):1837-46. doi: 10.1016/S0140-6736(16)00587-0. Epub 2016 Mar 10. PMID 26970723
- [Result] Spencer KR, Wang J, Silk AW, Ganesan S, Kaufman HL, Mehnert JM. Biomarkers for Immunotherapy: Current Developments and Challenges. Am Soc Clin Oncol Educ Book. 2016;35:e493-503. doi: 10.1200/EDBK_160766. PMID 27249758
- See also: Clinical Trial Facilitation Group. Recommendations related to contraception and pregnancy testing in clinical trials. Clinical Trial Facilitation Group. Recommendations related to contraception and pregnancy testing in clinical trials. 2014 — http://www.hma.eu/fileadmin/dateien/Human_Medicines/01-About_HMA/Working_Groups/CTFG/2014_09_HMA_CTFG_Contraception.pdf
- See also: Web page of the sponsor of the study — http://www.sogug.es/